CLINICAL TRIAL: NCT03173482
Title: Prevalence of Cesarean Section on Demand in Assiut University Hospital & Abnob Central Hospital
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, principal investigator, Assiut University
Other Study IDs: CSD
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Cesarean Section
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — asking about details of indication of cesarean section

SUMMARY:
Cesarean section on demand: defined as a primary cesarean section performed at the mother's request to avoid a vaginal birth, without any recognized medical or obstetric indication. The medical field now acknowledges a patient's right to actively participate in her choice of medical treatments, including method of delivery.

There are many reasons for a cesarean section on demand: fear of delivery, fear of pain, family pressure, a previous bad experience, more control over events, improved care, and maintaining the integrity of the pelvic floor. of the pelvic floor.

ELIGIBILITY:
Inclusion Criteria:

* Accepting to participate in the study.
* pregnant Women undergoing Cesarean section

Exclusion Criteria:

* pregnant Women undergoing Cesarean section due to medical or obstetric indication
* Caesarean hysterectomy .

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women attending the hospital for cesarean section
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
the percentage of cesarean section on request in patients | 1 year
  through a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No